CLINICAL TRIAL: NCT00945165
Title: Defining the Optimal Exercise Program to Improve Glycemic Control in Various Stages of Type 2 Diabetes.
Brief Title: Exercise and Glycemic Control in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-3-028
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia
Keywords: Continuous Glucose Monitoring System; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise intervention
- No exercise (Experimental)
  Interventions: Behavioral: No exercise

INTERVENTIONS:
Behavioral: Exercise intervention — various exercise characteristics
  Arms: Exercise
Behavioral: No exercise — No exercise control period
  Arms: No exercise

SUMMARY:
Hyperglycemia is an independent risk factor for the development of diabetic complications in type 2 diabetes. Exercise improves glycemic control, however, the role of exercise characteristics (e.g. intensity, type of exercise, timing, frequency) remains to be elucidated.

This study aims to assess the effect of several exercise characteristics on hyperglycemia in various subgroups of type 2 diabetes patiënts.

ELIGIBILITY:
Impaired glucose tolerant subjects

Inclusion Criteria:

* BMI 25 - 35 kg/m2
* Impaired Glucose Tolerant (according to ADA guidelines)

Exclusion Criteria:

* Cardiac disease (cardiac event in the last 5 years)
* Type 2 diabetes
* Use of orale blood glucose lowering medication or exogenous insulin
* HbA1c >10%

Insulin treated type 2 diabetes patients

Inclusion Criteria:

* BMI 25 - 35 kg/m2
* Insulin therapy
* diagnosed with type 2 diabetes >2 yr

Exclusion Criteria:

* Cardiac disease (cardiac event in the last 5 years)
* HbA1c >10%

Type 2 diabetes patients on oral blood glucose lowering medication

Inclusion Criteria:

* BMI 25 - 35 kg/m2
* diagnosed with type 2 diabetes >2 yr

Exclusion Criteria:

* Cardiac disease (cardiac event in the last 5 years)
* HbA1c >10%
* use of exogenous insulin

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-07; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Hyperglycemia | 24h

SECONDARY OUTCOMES:
Mean Blood Glucose | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem M van Dijk, MSc, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Klinkenberg LJ, van Dijk JW, Tan FE, van Loon LJ, van Dieijen-Visser MP, Meex SJ. Circulating cardiac troponin T exhibits a diurnal rhythm. J Am Coll Cardiol. 2014 May 6;63(17):1788-95. doi: 10.1016/j.jacc.2014.01.040. Epub 2014 Feb 26. PMID 24583293
- [Derived] van Dijk JW, Venema M, van Mechelen W, Stehouwer CD, Hartgens F, van Loon LJ. Effect of moderate-intensity exercise versus activities of daily living on 24-hour blood glucose homeostasis in male patients with type 2 diabetes. Diabetes Care. 2013 Nov;36(11):3448-53. doi: 10.2337/dc12-2620. Epub 2013 Sep 16. PMID 24041682
- [Derived] van Dijk JW, Tummers K, Stehouwer CD, Hartgens F, van Loon LJ. Exercise therapy in type 2 diabetes: is daily exercise required to optimize glycemic control? Diabetes Care. 2012 May;35(5):948-54. doi: 10.2337/dc11-2112. Epub 2012 Mar 7. PMID 22399700
- [Derived] van Dijk JW, Manders RJ, Tummers K, Bonomi AG, Stehouwer CD, Hartgens F, van Loon LJ. Both resistance- and endurance-type exercise reduce the prevalence of hyperglycaemia in individuals with impaired glucose tolerance and in insulin-treated and non-insulin-treated type 2 diabetic patients. Diabetologia. 2012 May;55(5):1273-82. doi: 10.1007/s00125-011-2380-5. Epub 2011 Nov 29. PMID 22124605
- See also: Website Muscle Metabolism Maastricht — http://www.m3-research.nl